CLINICAL TRIAL: NCT05835544
Title: Acute Responses to High-intensity Interval Exercise (HIIE) and Blood Flow Restriction (BFR)
Brief Title: Acute High Intensity Interval Training and Blood Flow Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Stephen Burns, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-2022-135
Record Dates: First submitted 2023-04-05; First posted 2023-04-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Activity, Motor
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIIT Control (Active Comparator): High intensity interval cycling
  Interventions: Other: Active Comparator: HIIT Control
- HIIT + BFR between cycling sets (Experimental): High intensity interval cycling with blood flow restriction applied between sets of cycling
  Interventions: Other: Experimental: HIIT + BFR between cycling sets
- HIIT + BFR moderate occlusion during cycling (Experimental): High intensity interval cycling with moderate blood flow restriction applied during cycling
  Interventions: Other: Experimental: HIIT + BFR moderate occlusion during cycling
- HIIT + BFR high occlusion during cycling (Experimental): High intensity interval cycling with high blood flow restriction applied during cycling
  Interventions: Other: Experimental: HIIT + BFR high occlusion during cycling

INTERVENTIONS:
Other: Active Comparator: HIIT Control — Complete 3 sets of five repetitions of 30 seconds cycling at 100% of maximal aerobic power with 30 seconds of active unloaded recovery between repetitions; 3 minutes of passive rest between sets.
  Arms: HIIT Control
Other: Experimental: HIIT + BFR between cycling sets — Complete 3 sets of five repetitions of 30 seconds cycling at 100% of maximal aerobic power with 30 seconds of active unloaded recovery between repetitions; 3 minutes of passive rest between sets. Blood flow restriction is applied for 2 minutes during the passive rest at 80% of limb occlusion pressure.
  Arms: HIIT + BFR between cycling sets
Other: Experimental: HIIT + BFR moderate occlusion during cycling — Complete 3 sets of five repetitions of 30 seconds cycling at 70% of maximal aerobic power with 30 seconds of active unloaded recovery between repetitions; 3 minutes of passive rest between sets. Blood flow restriction is applied during and between exercise repetitions at 50% of limb occlusion pressure and deflated during passive rest periods.
  Arms: HIIT + BFR moderate occlusion during cycling
Other: Experimental: HIIT + BFR high occlusion during cycling — Complete 3 sets of five repetitions of 30 seconds cycling at 70% of maximal aerobic power with 30 seconds of active unloaded recovery between repetitions; 3 minutes of passive rest between sets. Blood flow restriction is applied during and between exercise repetitions at 80% of limb occlusion pressure and deflated during passive rest periods.
  Arms: HIIT + BFR high occlusion during cycling

SUMMARY:
The study aims to look at the blood flow restriction (BFR) + high intensity interval training (HIIT) variables to induce an optimal acute training stimulus (i.e., acute responses in main outcome measures of muscular activation, muscular deoxygenation, and secondary outcome measures of heart rate (HR), blood lactate (bLa), subjective ratings of perceived exertion and discomfort)

The hypotheses for this study are: (i) BFR increases muscular deoxygenation, muscular activation when HIIT exercise is of the same intensity, (ii) however, comparing between a lower BFR + HIIT exercise intensity (e.g. 80% V̇O2max) and higher HIIT exercise intensity (e.g. 100% V̇O2max), muscular deoxygenation and activation will be similar but HR will be lower in the BFR + HIIT condition.

DETAILED DESCRIPTION:
This study revolves around the optimisation of blood flow restriction (BFR) and high-intensity interval training (HIIT) protocols for the racket sport athlete. The study aims to look at the BFR + HIIT variables to induce an optimal acute training stimulus. This can be achieved with the consideration of two main research questions: (i) What is the ideal combination of BFR cuff pressure and exercise intensity (i.e. cycling) to elicit favourable training stimuli, i.e., acute responses in main outcome measures of muscular activation, muscular deoxygenation, and secondary outcome measures of heart rate (HR), blood lactate (bLa), subjective ratings of perceived exertion and discomfort?; (ii) How does BFR + HIIT compare with traditional HIIT at a similar or higher exercise intensity in terms of these acute responses?

The hypotheses for this study are: (i) BFR increases muscular deoxygenation, muscular activation when HIIT exercise is of the same intensity, (ii) however, comparing between a lower BFR + HIIT exercise intensity (e.g. 80% V̇O2max) and higher HIIT exercise intensity (e.g. 100% V̇O2max), muscular deoxygenation and activation will be similar but HR will be lower in the BFR + HIIT condition.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age: 18-40 years
* Competed in competitive varsity sports (endurance, tennis, badminton, squash, football, basketball, etc.) at the varsity/club level
* Actively training for at least 2 sessions (1 - 1.5h) per week
* Healthy (free from illnesses) and no musculoskeletal injuries for the past 6 months
* No history of cardiometabolic, vascular diseases or similar conditions (high blood pressure, peripheral vascular diseases, heart diseases, metabolic syndrome, diabetes, stroke, etc.).
* Pass pre-participation health screening tests - Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) and Australian Institute of Sport (AIS) Blood Flow Restriction (BFR) pre-screening questionnaire (no history of any risk factors).
* Maximal oxygen uptake (VO2max) of ≥40mmol/min/kg during a maximal aerobic cycling test.
* Non-smoker
* Drink alcohol less than 3 times each week and less than 3 drinks each time

Exclusion Criteria:

* Any diagnosed form of cardiometabolic disease (CVD, diabetes, metabolic syndrome, hypertension)
* Any symptoms contraindication of exercise testing (eg chest pains)
* Any balance or dizziness problems
* Any chronic medical conditions (whether medicated or not)
* Any bone joint problems
* Any Physician diagnosed contraindications to exercise

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 24 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Heart rate | Measured and compared between each acute arm (condition)
  Heart rate using short-range telemetry
Blood lactate concentration | Measured and compared between each acute arm (condition)
  Fingertip capillary measure
Muscle activation | Measured and compared between each acute arm (condition)
  Surface electromyography of the vastus lateralis and biceps femoris muscles to determine electrical activity of the motor units (physiological parameter)
Muscle oxygenation | Measured and compared between each acute arm (condition)
  Near infra-red spectroscopy to examine regional tissue (the vastus lateralis muscle) oxygenation i.e, the percentage of haemoglobin and deoxyhaemoglobin (physiological parameter)

SECONDARY OUTCOMES:
Rating of perceived exertion | Measured and compared between each acute arm (condition)
  Borg Rating of Perceived Exertion scale 6-20 (6 = no exertion at all; 20 = maximal exertion)
Exertion and Pain scale | Measured and compared between each acute arm (condition)
  Borg Category-Ratio (CR) 10 scale (0 = No exertion at all; 10 = Maximal)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Burns, PhD, Principal Investigator — Nanyang Technological University
Locations (1):
- Human Bioenergetics Laboratory, National Institute of Education, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
All published data will be placed into the Data Repository of Nanyang Technological University National Institute of Education for public access upon publication.
Supporting Information: Analytic Code
Time Frame: Upon publication - permanent repository
Access Criteria: Public repository - exact web address available upon publication.
URL: http://researchdata.nie.edu.sg/

REFERENCES:
- [Derived] Chua M, Sim A, Burns SF. Acute physiological and perceptual responses to three blood flow restricted interval exercise protocols: a randomised controlled trial. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-13. doi: 10.1139/apnm-2024-0423. PMID 39919270